CLINICAL TRIAL: NCT03530410
Title: Gastric and Autonomic Functions in Patients With Intragastric Balloon
Status: Withdrawn | Type: Observational
Why Stopped: The study did not recruit any participant.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00154036
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Obesity, Morbid
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with intragastric balloon: Patients who will receive an intragastric balloon placement for weight loss
  Interventions: Device: Intragastric balloon placement

INTERVENTIONS:
Device: Intragastric balloon placement — Patients will have endoscopic placement of intragastric balloon that will be removed endoscopically after 6 months

SUMMARY:
The study aims to measure the effect of intragastric balloon on gastric function, particularly gastric accommodation and pace making, and the possible underlying changes in autonomic function

DETAILED DESCRIPTION:
The intragastric balloon is a space-occupying device that is hypothesized to function by inducing early satiety. Additionally, insertion of an intragastric balloon causes delayed gastric emptying; longer gastric emptying times after balloon insertion are correlated with more weight loss. The exact mechanism of function, however, is not clear and likely multifactorial. The investigators hypothesize that the intragastric balloon causes weight loss by affecting gastric and autonomic function, including pace-making and accommodation, and that the difference in responsiveness among patients may be mediated by differences in gastric function.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo intragastric balloon implantation
* Ability to comply to study schedule.

Exclusion Criteria:

* Unable to give informed consent
* Currently taking prokinetic, anticholinergic or dopaminergic agents which could potentially modify gastric motility
* Have a history of bariatric or gastrointestinal surgery
* Pregnant or preparing to conceive a child.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo intragastric balloon implantation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Gastric slow waves | 1 year
  A noninvasive method similar to electrocardiography, called electrogastrography, will be used in this study to assess the effects of intragastric balloon on gastric slow waves
Gastric accommodation | 1 year
  A noninvasive nutrient drink test will be performed and accommodation will be assessed using a symptom (fullness, nausea, belching of air, cramps in the abdomen, bloating, and pain) scale 0 to 3 points with higher values indicating more and/or greater symptoms
Autonomic function | 1 year
  The ECG will be recorded simultaneously with the Electrogastrograph (EGG) and will be used to noninvasively assess the vagal and sympathetic activities as well as the sympathovagal ratio

SECONDARY OUTCOMES:
Gastroparesis cardinal symptom index (GCSI) questionnaire | 1 year
  Gastroparesis symptoms questionnaire. Score ranges from 0 (none) to 45 (very severe)
Gastroesophageal reflux disease-health related quality of life (GERD-HRQL) questionnaire | 1 year
  A tool for measuring symptom severity in gastroesophageal reflux disease (GERD). Score ranges from 0 (no symptoms) to 75 (worst symptoms)
Dyspepsia symptom severity index (DSSI) questionnaire | 1 year
  A tool for assessing the severity of symptoms commonly associated with dyspepsia. Score ranges from 0 to 4 based on severity.
SF-36 Questionnaire | 1 year
  36 item questionnaire which measures Quality of Life (QoL) across eight domains. Scores range from 0% (lowest level of functioning) to 100% (highest level of functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Kumbhari, MD, Principal Investigator — Johns Hopkins University